CLINICAL TRIAL: NCT03591523
Title: Blood Flow Measurement in Cervical and Cerebral Arteries Using Quantitative Magnetic Resonance Angiography and Cervical and Transcranial Duplex Sonography
Brief Title: Blood Flow Measurement Using Quantitative Magnetic Resonance Angiography and Duplex Sonography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Palacky University (Other)
Collaborators: České Budějovice Hospital (Other)
Responsible Party: Principal Investigator, Ing. Irena Jedličková, Study Manager, Palacky University
Other Study IDs: 28042018
Record Dates: First submitted 2018-07-07; First posted 2018-07-19 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Cerebrovascular Circulation
Keywords: cerebrovascular circulation; arterial blood flow; magnetic resonance; duplex sonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspicion of vascular pathology: Subjects indicated to quantitative MR angiography and duplex sonography for suspicion of cervical or intracranial vascular pathology
  Interventions: Diagnostic Test: Quantitative MR angiography; Diagnostic Test: Duplex sonography

INTERVENTIONS:
Diagnostic Test: Quantitative MR angiography — Quantitative MR angiography: A standard axial 3-dimensional time-of-flight (TOF) MRA of intracranial and cervical arteries will be obtained. Then, the acquired images will be transmitted to the workstation to reconstruct 3D surface-rendered vessel images. After determining optimal perpendicular scan plane and setting the baseline coordinates , retrospectively gated, fast 2-dimensional phase-contrast sequence will be performed. Velocity encoding will be automatically adjusted by NOVA software.
  Other Names: qMRA
Diagnostic Test: Duplex sonography — Duplex sonography of cervical arteries will be performed using 5 - 12 MHz linear duplex probe and transcranial color-coded duplex sonography will be performed using 2 - 5 MHz transcranial duplex probe. Peak systolic velocity, end diastolic celocity, mean blood flow velocity and arterial diameter will be measured with automatic calculation of blood flow velocity in each arterial segment.
  Other Names: DS

SUMMARY:
The aim of the study is to assess the correlation of blood flow measurement in cervical and intracranial arteries between quantitative magnetic resonance angiography (qMRA) and duplex sonography (DS) and inter-/intra-investigators reliability of both methods in common clinical practice. A total of 21 subjects indicated to qMRA or DS for suspicion of cervical or intracranial vascular pathology will be included. All patients will undergo qMRA and DS of the cervical and intracranial arteries with measurement of blood flow in bilateral common carotid artery (CCA), internal carotid artery in proximal part distally to carotid bulb (ICA) and in distal carotid siphon (ICA-siphon), external carotid artery (ECA), vertebral artery in V2 (V2-VA) and V4 (V4-VA) segments, middle cerebral artery (MCA), anterior cerebral artery in pre-communicant (ACA1) and post-communicant (ACA2) part, posterior cerebral artery in pre-communicant (PCA1) and post-communicant (PCA2) part and basilar artery (BA) the cerebral artery. Correlations between measurements will be evaluated using Spearman's correlation coefficient or kappa coefficient and inter-class correlation coefficient (ICC).

DETAILED DESCRIPTION:
Introduction: Measurement of blood flow in cervical and cerebral arteries is important not only for accurate diagnosis of neurovascular diseases but also for refinement of the indication of invasive treatment. Quantitative MR angiography (qMRA) with NOVA flow analysis system and duplex sonography (DS; duplex sonography of cervical arteries and transcranial color-coded duplex sonography) are non-invasive diagnostics methods which could be used for measurement of blood flow in cervical and intracranial arteries.

Aim: The aim of the study is to assess the correlation of blood flow measurement in cervical and intracranial arteries between qMRA and DS in common clinical practice. The secondary aims are to assess the inter-investigator and intra-investigator correlations of both qMRA and DS in blood flow measurement.

Methods: A total of 21 subjects indicated to qMRA or DS for suspicion of cervical or intracranial vascular pathology will be included.

Inclusion criteria: male or female; age 25 - 70 years; signed informed consent. Exclusion criteria: contraindication to magnetic resonance; uncontrolled involuntary movements; other condition preventing long-term quiet lying.

All patients will undergo qMRA and DS of the cervical and intracranial arteries within 2 hours. The NOVA flow analysis system will calculate blood flow in individual segments. In DS, angle corrected blood flow velocities (peak systolic velocity - PSV, end-diastolic velocity - EDV, mean velocity - Vmean) will be measured in individual segments with measurement of arterial in the B-Mode or Color Mode with automatic calculation of blood flow.

The blood flow will be assessed in the following arterial segments: bilateral common carotid artery (CCA), internal carotid artery in proximal part distally to carotid bulb (ICA) and in distal carotid siphon (ICA-siphon), external carotid artery (ECA), vertebral artery in V2 (V2-VA) and V4 (V4-VA) segments, middle cerebral artery (MCA), anterior cerebral artery in pre-communicant (ACA1) and post-communicant (ACA2) part, posterior cerebral artery in pre-communicant (PCA1) and post-communicant (PCA2) part and basilar artery (BA) the cerebral artery.

At least 2 patients will undergo qMRA and DS performed by the same investigators twice in the time interval of 2 - 10 days and DS will be performed in all patients by 2 sonographers using 2 different machines for assessment of inter-investigator and intra-investigator reliability.

All investigators will be blinded to the diagnosis and measurement performed using other diagnostics method.

In all patients will be collecting following data: blood pressure, weight, height, age, gender, time of examination Statistics: Correlations between measurements will be evaluated using Spearman's correlation coefficient or kappa coefficient and inter-class correlation coefficient (ICC).

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age 25 - 70 years
* suspicion of cervical or intracranial vascular pathology
* signed informed consent.

Exclusion Criteria:

* contraindication to magnetic resonance
* uncontrolled involuntary movements
* other condition preventing long-term quiet lying.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects indicated to qMRA or DS for suspicion of cervical or intracranial vascular pathology will be included
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Blood flow measurement | 6 weeks
  Correlation of blood flow measurement between qMRA and DS

SECONDARY OUTCOMES:
Intra-investigator reliability of quantitative magnetic resonance angiography | 6 weeks
  Intrainvestigator reliability of blood flow measurement using qMRA performed by the same investigators in two sessions
Inter-investigator reliability of duplex sonography | 6 weeks
  Inter-investigator reliability of blood flow measurement using duplex sonography performed by 2 investigators
Intra-investigator reliability of duplex sonography | 6 weeks
  Intra-investigator reliability of blood flow measurement using duplex sonography performed by the same investigator in two sessions

CONTACTS AND LOCATIONS:
Overall Officials: David Skoloudik, Prof. Dr., Principal Investigator — Palacký University Olomouc, Center for Science and Research
Locations (1):
- Nemocnice Ceske Budejovice, České Budějovice, Czechia

IPD SHARING:
Plan to Share IPD: Undecided